CLINICAL TRIAL: NCT00531401
Title: Salirasib for Treatment of Advanced Non-Small Cell Lung Cancer: a Phase II Study
Brief Title: Study of Salirasib to Treat Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concordia Pharmaceuticals, Inc (Industry)
Responsible Party: Victor Bauer, Concordia Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCA-FTS-201
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — farnesylthiosalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Salirasib — 600mg BID until disease progression or unacceptable toxicity occurs.

SUMMARY:
The purpose of this study is to determine whether Salirasib is effective to shrink or prevent the growth of the tumors associated with non-small cell lung cancer in both patients who are newly diagnosed or have recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Non-Small Cell Lung Cancer not amenable to curative therapy with surgery or radiation
* Measurable disease
* Adenocarinoma of the lung, have not received prior chemotherapy for the malignancy and has a ≥ 15 pack year history of smoking; OR previously treated with recurrent disease and documented KRAS mutation
* Last dose of radiotherapy > 3 weeks prior to study entry and recovered from all acute toxicities associated with the prior therapy
* No history of another malignancy in the past 5 years except treated non-melanomatous skin cancer or superficial bladder cancer or carcinoma-in-situ of the cervix
* Karnofsky Performance status of 70 or greater
* Body Weight > 50 kg
* Life expectancy ≥ 3 months
* Serum Creatinine ≤2.0 mg/dL, total bilirubin ≤ 2.0 mg/dL, ALT and AST ≤ 3x ULN, alkaline phosphatase ≤ 5x ULN, WBC > 3000/mm³, ANC ≥ 1500/mm³, platelets ≥ 100,000/mm³, hemoglobin ≥ 10g/dL.
* No coexisting cardiac or medical problems that would limit compliance in the study
* Willing to undergo blood sampling for pharmacokinetic analysis
* Negative pregnancy test, if applicable

Exclusion Criteria:

* Evidence of active heart disease including myocardial infarction within previous 3 months
* Active infectious process
* Active central nervous system metastases (requiring increasing doses of corticosteroids over the prior month, known progressing lesions)
* Pregnant or lactating
* Major surgery without full recovery or major surgery within 3 weeks prior to treatment start
* QTc Interval > 470 msec
* Gastrointestinal tract disease resulting in inability to take or absorb oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Rate of non-progression (as reflected in the tumor control rate of percent patients with CR+PR+SD) defined as the number of patients whose tumor did not progress (<20% tumor increase to total disappearance of tumor according to RECIST) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Riely, MD PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States